CLINICAL TRIAL: NCT01862523
Title: Unraveling the Mechanisms of Capsaicin Treatment in Idiopathic Rhinitis Patients and Controls by Measuring Mucosal Potentials in the Nose.
Brief Title: Mechanisms of Capsaicin Treatment in Idiopathic Rhinitis Patients and Controls
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mucosal potentials in the nose
Record Dates: First submitted 2012-09-05; First posted 2013-05-24 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- diluent (Placebo Comparator): diluent
  Interventions: Biological: diluent
- capsaicin (Experimental): capsaicin
  Interventions: Biological: Capsaicin
- control healthy volunteers (No Intervention): control healthy volunteers

INTERVENTIONS:
Biological: Capsaicin — Thirty-three* well-characterized IR patients will be recruited and screened for participation in this study with nasal capsaicin spray (0,1 mmol/l ) using the treatment regimen described by van Rijswijk et al. (1 x 5 applications in one day, with 1 hour between each application)
  Arms: capsaicin
Biological: diluent — diluent
  Arms: diluent

SUMMARY:
Capsaicin nasal spray is used in daily practice against IR without knowledge about the exact mechanisms involved in this treatment. Therefore, this study aims to address this issue by studying the functional (electrophysiologic) changes after specific stimulations in IR patients and healthy controls before and after capsaicin/placebo treatment.

DETAILED DESCRIPTION:
As an essential step towards the improvement of the treatment of IR we will investigate the neural mechanisms underlying the therapeutic action of capsaicin. In particular, we plan to evaluate the effects of capsaicin on the functional properties of the innervation of nasal mucosa by monitoring the trigeminal nerve activity using measurements of negative mucosa potentials (NMP). NMPs, will be evoked by chemical and thermal stimuli in IR patients and healthy controls. Considering the evidence suggesting a role of sensory C-fibers in the pathophysiology of IR, we will employ low concentrations of irritants that specifically activate receptors expressed in those fibers, i.e., capsaicin for TRPV1 and cinnamaldehyde and allyl-isothiocyanate (mustard oil) for TRPA1. The same stimulations will be performed immediately after capsaicin treatment, and after 4 weeks, 3 months and 6 months. This will allow for an objective assessment of the functionality of the C-fiber innervation before the treatment, during the phase of therapeutic response and during the period of recurrence of the IR symptoms. The results of the NMP measurements will be contrasted with the therapeutic response and with evaluations of nasal congestion, nasal sensitivity and the presence of neuro-mediators found in nasal biopsies. Importantly, the independent assessment of the NMP responses mediated by either TRPV1 or TRPA1 will allow determining the specific role of these nociceptors in the pathophysiology of IR, which, in turn, may help to design more specific and effective therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent (> 52w) rhinological symptoms: nasal discharge, sneezing, congestion for an average of at least 1 h per day for at least 5 days during a period of 14 days, negative skin prick test or negative RAST, and without structural abnormalities explaining nasal obstruction will be proposed to participate in the trial.
2. Age > 18 and < 60 years
3. Written informed consent
4. Willingness to adhere to visit schedules
5. Adequate contraceptive precautions in female patients with childbearing potential
6. Unresponsiveness to nasal steroid spray (4 weeks of use)

Exclusion Criteria:

1. Age < 18 and > 60 years
2. Patients with AR, demonstrated by either positive skin prick test or RAST
3. Asthma
4. Structural abnormalities: nasal polyps, severe septal deviation (septum reaching concha inferior or lateral nasal wall.
5. Systemic steroid treatment less than 4 weeks before the inclusion in the study.
6. Nasal steroid spray less than 4 weeks before the inclusion, oral leukotriene antagonists or long-acting antihistamines less than 2 weeks before the inclusion.
7. Inability of the patient to stop taking medication affecting nasal function.
8. Evidence of infectious rhinitis/rhinosinusitis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
negative mucosa potentials | baseline, 1, 3 and 6 months
  change in negative mucosa potentials (baseline vs 1, 3 and 6 months after treatment)by measurement of AUC, delay-time and amplitude

SECONDARY OUTCOMES:
visual analogue scale | baseline, 1, 3 and 6 months
  change of visual analogue scale of the administered stimuli (baseline vs 1, 3 and 6 months after treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Van Gerven, Doctor, Principal Investigator — UZ Leuven; Peter Hellings, Doctor, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium